CLINICAL TRIAL: NCT06258967
Title: A Prospective Randomized Controlled Trail of Ciprofol Titrated Induction in Reducing Post-induction Hypotension in Geriatric Patients Under General Anesthesia
Brief Title: Ciprofol Titrated Induction in Reducing Post-induction Hypotension in Geriatric Patients
Acronym: CTIH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2023ZSLYEC-636
Record Dates: First submitted 2024-01-04; First posted 2024-02-14 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-01

CONDITIONS: Post Induction Hypotension; Elderly
MeSH Terms: interventions — (2-(1R)-1-cyclopropyl)ethyl-6-isopropyl-phenol; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propofol (Active Comparator): Propofol is administered at a rate of 15mg/kg*h for patient induction. After 60 seconds, a sedation assessment is initiated until the patient loses consciousness.Then adjust the propofol dose to 5mg/kg/h and make further dose adjustments based on the patient's response and BIS value, with increments or decrements ranging from 1mg/kg/h, within a total range of 3-8mg/kg/h.
  Interventions: Drug: propofol
- Ciprofol (Experimental): Cprofol is administered at a rate of 3mg/kg*h for patient induction. After 60 seconds, a sedation assessment is initiated until the patient loses consciousness.Then adjust the propofol dose to 1mg/kg/h and make further dose adjustments based on the patient's response, with increments or decrements ranging from 0.2mg/kg/h, within a total range of 0.6-1.6mg/kg/h.
  Interventions: Drug: ciprofol

INTERVENTIONS:
Drug: ciprofol — Patients receive ciprofol as general anesthesia induction drug, using the titrated anesthesia method.
  Arms: Ciprofol
Drug: propofol — Patients receive propofol as general anesthesia induction drug, using the titrated anesthesia method.
  Arms: Propofol

SUMMARY:
Geriatric patients undergoing general anesthesia face a significant challenge, with the induction phase contributing to 50% of hypotensive events.

Titrated anesthesia, involving gradual drug administration, suits elderly induction. However, propofol in titrated anesthesia tends to induce hypotension. In contrast, Ciprofol (HSK3486), a novel anesthetic, reduces hypotension during induction. This study compares hypotension incidences during induction and post-induction phases, agitation rates during recovery, perioperative awareness, postoperative delirium, and parameters in elderly patients induced with Ciprofol versus propofol through titrated anesthesia. The goal is to clarify a medically optimized anesthesia protocol for elderly patients during titrated anesthesia induction in general anesthesia.

DETAILED DESCRIPTION:
As the global population ages, there is a growing demand for surgical interventions among the elderly. However, this demographic is concurrently faced with an increased susceptibility to postoperative complications. Notably, the geriatric population undergoing general anesthesia exhibits a higher incidence of hypotension, intricately linked with a spectrum of postoperative issues. The induction phase of general anesthesia, constituting 50% of hypotensive events, presents a significant challenge in mitigating hypotension.

Titrated anesthesia, characterized by gradual and individualized drug administration, emerges as a suitable approach for the induction of general anesthesia in the elderly. Nevertheless, the administration of propofol through titrated anesthesia maintains an observable tendency to induce hypotension.

In contrast, Ciprofol (HSK3486), a novel anesthetic agent, demonstrates a reduced propensity for precipitating hypotension during the induction of anesthesia. This investigative study aims to meticulously examine and compare the incidences of hypotension during both the induction and post-induction phases. Furthermore, it endeavors to delineate differences in the rates of agitation during the recovery phase, perioperative awareness, postoperative delirium, and other relevant parameters among elderly patients induced with ciprofol versus propofol via titrated anesthesia.

A sample size of 80 patients in each group will be selected by a prior power analysis on the basis of the following assumptions: (1) the rate of hypotension in group Propofol was 57%; and 30%in group Cipropfol (2)α=0.05, (4) power 90% and .(5) missed follow-up rate 12%.

After obtaining informed consent, all participants will be randomized to one of the trial groups using a stratified method. A 20G catheter will be inserted into the radial artery before anesthesia induction. Vital signs will be recorded from 3 minutes before general induction until 15 minutes after tracheal intubation. Participants in Group P will undergo induction with propofol, starting at a rate of 15mg/kg/h until loss of consciousness, followed by an adjustment to a slower infusion rate. In contrast, Group C will receive ciprofol at a rate of 3mg/kg/h. Following the intervention period, all participants will receive sevoflurane and remifentanil until the conclusion of the surgery. Both groups will be followed up for 7 days postoperatively to assess perioperative awareness, postoperative delirium, quality of recovery, and postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years and age < 90 years.
* ASA (American Society of Anesthesiologists) physical status classification 1-3.
* Scheduled for elective general anesthesia surgery.

Exclusion Criteria:

* Participants already enrolled in other studies or those already assigned in this study .
* BMI (Body Mass Index) ≤ 18 or ≥ 30 kg/m2.
* Preoperative assessment indicating a challenging airway or a risk of aspiration, requiring a slow induction for intubation.
* Presence of severe liver or kidney disease (GFR ≤ 30 ml/min/1.73m2 or requiring renal replacement therapy; Child-Pugh class C for liver function).
* Patients with severe uncontrolled hypertension (preoperative SBP ≥ 180 mmHg or DBP ≥ 110 mmHg).
* Individuals with arrhythmias and severe valvular diseases, including high-degree atrioventricular block (Mobitz type II or third-degree block); symptomatic bradycardia; symptomatic ventricular arrhythmias; prolonged Q-T interval; supraventricular arrhythmias combined with an uncontrolled ventricular rate > 100 bpm (at rest); new-onset ventricular tachycardia; uncontrolled atrial fibrillation (ventricular rate ≥ 110 bpm); atrial flutter; severe aortic valve stenosis (mean pressure gradient > 40 mmHg; valve area < 1 cm2; symptomatic); severe mitral valve stenosis (progressive breathlessness during exertion; exertional syncope; heart failure).
* Patients diagnosed with schizophrenia, epilepsy, Parkinson's disease, severe cognitive impairment, intellectual disability, hearing impairment.
* Individuals with a history of alcoholism or long-term use of sedatives and analgesics.
* Previous allergic reactions to medications used in this study.
* Individuals already under vasoconstrictor treatment before anesthesia induction.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2024-12-24 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The difference in the incidence of hypotension occurring 15 minutes after successful intubation between the two groups. | From successful tracheal intubation to 15 minutes later.
  Hypotension is defined as a mean arterial pressure (MAP) of 65 mmHg or lower. The occurrence of hypotension in each group will be documented.

SECONDARY OUTCOMES:
Time-weighted area under the curve of blood pressure during the post-induction phases of anesthesia with a mean arterial pressure (MAP) < 65 mmHg. | From successful tracheal intubation to 15 minutes later.
  This outcome will be caculated as: (65-MAP)(mmHg)*Time(min)
Time-weighted area under the curve of blood pressure during the induction and post-induction phases of anesthesia with a mean arterial pressure (MAP) ≤ 70% of the baseline value. | From successful tracheal intubation to 15 minutes later.
  This outcome will be caculated as: (70%*MAPbaseline -MAP)(mmHg)*Time(min)
Time-weighted area between the curve of blood pressure and the target MAP(110mmHg,120mmHg) during the post-induction period | From successful tracheal intubation to 15 minutes later.
  This outcome will be caculated as: (MAP-110)(mmHg)*Time(min) and (MAP-110)(mmHg)*Time(min) and (MAP-120)(mmHg)*Time(min)
The dose of norepinephrine used during the induction and post-induction periods. | From the administration of general anesthesia with an induction drug to 15 minutes after tracheal intubation has been completed.
  Norepinephrine dosage in each group will be recorded.
Total time for patient loss of consciousness | During anesthesia induction
  Time from anesthetic drug adminisered to patient's OAA/S score reached 1
Trends in CO( cardiac output) | from 1min before aneshesia induction until 20minuts after study durg administered.
  A divice will analyse the invasive BP wave ,caculated patient's CO, and will be recorded.
Incidence of agitation during the post-anesthesia recovery period and early postoperative delirium . | 30min and 1hour after patients arrived the PACU
  Patients will be astimated using the Richmond Agitation Sedation Scale (RASS, the score between -5~+4) and Confusion Assessment Method for the Intensive Care Unit (CAM-ICU).The rate of agitation of each group will be recorded.
Incidence of perioperative awareness | 1,2,3 days postoperatively
  The rate of awareness in each group will be recorded.
Incidence of postoperative nausea and vomiting | postoperative 1,2,3days
  Rate of participants with nausea and vomiting
Incidence of Postoperative delirium | 1,2,3days postoperatively
  The postoperative delirium will be screened using the 3-Minute Diagnostic confusion assessment method (3D-CAM).If patients is in the ICU ,then will be screened with CAM-ICU method.The rate of deilirium in each group will be recorded.
Incidence of complications within 7 days postoperatively. | 7 days postoperatively.
  All complications were evaluated according to the Clavian-Dindo Classification of Surgical Complications (CD). The CD scoring system is divided into five levels, with the more severe the complication, the higher the score.The occurrence of Clavien-Dindo grade ≥2 in each group will be recorded.
The difference of Postoperative Quality of Recovery-15 (QoR-15) score. | 1,2,3 days postoperatively
  The Quality of Recovery-15 (QoR-15) score,which has a max score of 150,and minimum score of 0, and a higher score means a bettery recovery. The score of each group will be recorded.
Time-weighted area under the curve of blood pressure during the post-induction phases of anesthesia with a mean arterial pressure (MAP) <55 mmHg. | From successful tracheal intubation to 15 minutes later.
  This outcome will be caculated as: (55-MAP)(mmHg)*Time(min)
Time-weighted area upon the curve of blood pressure during the post-induction phases of anesthesia with a mean arterial pressure (MAP) ≥140 mmHg. | From successful tracheal intubation to 15 minutes later.
  This outcome will be caculated as: (MAP-140)(mmHg)*Time(min)
Time-weighted area upon the curve of blood pressure during the post-induction phases of anesthesia with a mean arterial pressure (MAP) >110 mmHg. | From successful tracheal intubation to 15 minutes later.
  This outcome will be caculated as: (MAP-110)(mmHg)*Time(min)
Time-weighted area upon the curve of blood pressure during the post-induction phases of anesthesia with a mean arterial pressure (MAP) >120 mmHg. | From successful tracheal intubation to 15 minutes later.
  This outcome will be caculated as: (MAP-120)(mmHg)*Time(min)

CONTACTS AND LOCATIONS:
Locations (1):
- the Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China